CLINICAL TRIAL: NCT00166530
Title: A Prospective Randomized Open Label Blinded Endpoint Multicenter Study in Patients With Coronary Artery Disease to Assess the LDL Lowering Effect of Switching to Ezetimibe (+) Simvastatin for Cholesterol Lowering, Compared the Dose of the Statin Used.
Brief Title: EASEGO Study: Doubling of Atorvastatin/Simvastatin or INEGY in Patients With Hypercholesterolemia and Coronary Artery Disease(CAD)(0653A-089)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-089; MK0653A-089; 2005_059
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin; Atorvastatin

ARMS (2):
- 1 (Active Comparator): Arm 1: Active comparator
  Interventions: Drug: simvastatin; Drug: atorvastatin
- 2 (Experimental): Arm 2: Drug
  Interventions: Drug: ezetimibe (+) simvastatin

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Vytorin® combination tablet of ezetimibe 10 mg plus simvastatin 20 mg once daily for 12 weeks. Tablets
  Other Names: MK0653A; Vytorin®; INEGY™
  Arms: 2
Drug: simvastatin — Zocor®; simvastatin 40 mg once daily for 12 weeks. Tablets
  Other Names: MK0733; Zocor®
  Arms: 1
Drug: atorvastatin — 20 mg atorvastatin once daily for 12 weeks. Tablets
  Arms: 1

SUMMARY:
In patients with coronary artery disease and a LDL-C level between 2.5 mmol/L and 5.0 mmol/L on a stable (> 4 weeks) statin starting dose (simvastatin 20 mg or atorvastatin 10 mg), investigate what the LCL-C lowering efficacy is of doubling the statin dose (to 40 mg simvastatin or 20 mg atorvastatin) versus a combination tablet of ezetimibe 10 mg plus simvastatin 20 mg once daily for 12 weeks. It is postulated that more patients reach their LDL-C treatment goal with the combination tablet compared to doubling the starting dose. Furthermore, the effect of both treatment regimens on other lipid parameters, safety and LDL-subfractions will be measured.

DETAILED DESCRIPTION:
Patients with simvastatin 20 mg or atorvastatin 10 mg were randomized to (1) double statin dose (to 40 mg simvastatin or 20 mg atorvastatin) or (2) switch to a combination tablet of ezetimibe 10 mg plus simvastatin 20 mg once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female 18 years of age.
* Patient is on a stable daily statin starting dose for the past 4 weeks of either: atorvastatin 10 mg or; simvastatin 20 mg
* lipid values while on statin monotherapy treatment: LDL-C level of > 2.5 mmol/L to * 5.0 mmol/L, triglycerides < 4.0 mmol/L and total cholesterol < 7.0 mmol/L.
* Patient with established coronary artery disease such as stable angina; history of myocardial infarction; history of percutaneous coronary intervention (PTCA with or without stent placement); coronary stenosis on angiography; history of unstable angina or non-Q wave myocardial infarction; history of coronary artery bypass graft surgery (CABG); positive MIBI scan. Patients have to be in a stable medical condition.

Exclusion Criteria:

* Patients in whom cholesterol lowering medication regime has changed in the previous 4 weeks.
* Patients who have been treated with any other investigational drug within 3 months of Visit 1.
* Patients who are pregnant or lactating.
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the patient or interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Switching to a combination tablet of ezetimibe 10 mg plus simvastatin 20 mg is superior to doubling the statin dose as demonstrated by the percentage of patients reaching goal after 12 weeks of treatment. | after 12 weeks of treatment

SECONDARY OUTCOMES:
Switching to a combination tablet of ezetimibe 10 mg plus simvastatin 20 mg will lower LDL-C more than doubling the statin dose as demonstrated by the percentage change from treated baseline in total and LDL-cholesterol after 12 weeks of treatment. | after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Roeters van Lennep HW, Liem AH, Dunselman PH, Dallinga-Thie GM, Zwinderman AH, Jukema JW. The efficacy of statin monotherapy uptitration versus switching to ezetimibe/simvastatin: results of the EASEGO study. Curr Med Res Opin. 2008 Mar;24(3):685-94. doi: 10.1185/030079908X273273. Epub 2008 Jan 25. PMID 18226326
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html